CLINICAL TRIAL: NCT00497289
Title: Double-blind, Prospective, Randomized Comparison of a Medium Chain Triglycerides (MCT)/Long Chain Triglycerides (LCT)/Fish Oil (FO) Containing 20% Lipid Emulsion With a MCT/LCT Emulsion (20%) for Parenteral Nutrition in Preterm Infants
Brief Title: Comparison of Two Different Lipid Emulsions for Parenteral Nutrition in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HC-G-H-0404
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Preterm Infants; Parenteral Nutrition n-3 Fatty Acids
Keywords: n-3 Polyunsaturated Fatty Acids (PUFA); parenteral nutrition; preterm infant
MeSH Terms: conditions — Hyperphagia; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lipidem 20 %
  Interventions: Drug: Lipidem 20%
- 2 (Active Comparator): Lipofundin MCT/LCT 20%
  Interventions: Drug: Lipofundin MCT/LCT 20 %

INTERVENTIONS:
Drug: Lipofundin MCT/LCT 20 % — daily i.v. infusion for up to 5 days
  Arms: 2
Drug: Lipidem 20% — daily i.v. infusion for up to 5 days
  Arms: 1

SUMMARY:
The study shall provide evidence for the save and efficient use of a fish oil containing lipid emulsion in parenteral nutrition of preterm infants.Safety will be assessed by monitoring hepatological and hematological laboratory parameters. Efficiency will be assessed by monitoring of inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* prematurity (birth weight 500 - 1500 g)
* postnatal age <= 72 h
* need for cumulative parenteral energy supply of at least 70% during study duration
* signed informed consent form

Exclusion Criteria:

* simultaneous participation in another clinical study
* platelet count below 50000 /ml
* cumulative enteral energy supply of > 30 % during study duration
* serious congenital infections and/or diseases
* serious metabolic disturbances
* severe cranial bleeding (Papile III, IV)
* need for administration of blood products
* contra-indication for iv lipid administration
* withdrawal of consent

Ages: 5 Hours to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold V. Koletzko, Prof., MD, Principal Investigator — Dr. von Hauner Children´s Hospital, University of Munich
Locations (2):
- Germany (2):
  - Neonatology of the Pediatric University Hospital, Munich, Bavaria
  - Ernst Moritz Arndt University , Childrens Hospital, Greifswald

RESULTS

PARTICIPANT FLOW:
Groups:
- Lipidem 20 %: Lipidem 20 %
  Lipidem 20%: daily i.v. infusion for up to 5 days
- Lipofundin MCT/LCT 20%: Lipofundin MCT/LCT 20%
  Lipofundin MCT/LCT 20 %: daily i.v. infusion for up to 5 days
Period: Overall Study
Arm/Group | Lipidem 20 % | Lipofundin MCT/LCT 20%
Started | 24 | 24
Completed | 19 | 18
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- MCT:LCT:FO / 5:4:1: Lipidem 20%: daily i.v. infusion for up to 5 days
- MCT:LCT / 1:1: Lipofundin MCT/LCT 20 %: daily i.v. infusion for up to 5 days
- Total: Total of all reporting groups
Arm/Group | MCT:LCT:FO / 5:4:1 | MCT:LCT / 1:1 | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: hours] | 12.38 (19.38) | 13.74 (21.89) | 13.06 (20.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Germany | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Safety: Alanine Transaminase (ALT)
Description: Change in ALT between pre/post treatment
Time Frame: on Study day -1 & 6
Population: A duration of treatment with study medication over less than 6 days was regarded as the only major deviation from the protocol. Therefore all available values were used for analysis.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MCT:LCT:FO / 5:4:1 | MCT:LCT / 1:1
Number analyzed (Participants) | 15 | 19
U/L | -0.83 (4.61) | -3.27 (7.81)
Statistical Analysis 1: Comparison: MCT:LCT:FO / 5:4:1 vs MCT:LCT / 1:1; Test type: Superiority; p = 0.3654, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Efficacy: Interleukin-6 (IL-6)
Description: Change of IL-6 Measurement pre/post treatment
Time Frame: on Study day -1 & 6
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- MCT:LCT:FO / 5:4:1: Lipidem 20 %
  Lipidem 20%: daily i.v. infusion for up to 5 days
- MCT:LCT / 1:1: Lipofundin MCT/LCT 20%
  Lipofundin MCT/LCT 20 %: daily i.v. infusion for up to 5 days
Arm/Group | MCT:LCT:FO / 5:4:1 | MCT:LCT / 1:1
Number analyzed (Participants) | 19 | 17
pg/mL | -42.23 (197.10) | -68.74 (101.67)
Statistical Analysis 1: Comparison: MCT:LCT:FO / 5:4:1 vs MCT:LCT / 1:1; Test type: Superiority; p = 0.0264, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From enrolment into study at least 6 days or longer if medically indicated.
Groups:
- MCT/LCT/FO-containing 20% Fat Emulsion: Preterm infants received a study treatment by parenteral route with MCT/LCT/FO
  Lipidem 20%: daily i.v. infusion for up to 6 days
- MCT/LCT Emulsion (20%): Preterm infants received a study treatment by parenteral route with MCT/LCT
  Lipofundin MCT/LCT 20 %: daily i.v. infusion for up to 6 days
Arm/Group | MCT/LCT/FO-containing 20% Fat Emulsion | MCT/LCT Emulsion (20%)
Serious Adverse Events (participants affected / at risk) | 22/24 | 19/24
Other Adverse Events (participants affected / at risk) | 24/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCT/LCT/FO-containing 20% Fat Emulsion (N=24) | MCT/LCT Emulsion (20%) (N=24)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Neonatal infection (Infections and infestations) | 1 (1) | 0 (0)
Amniotic infection syndrome of Blane (Infections and infestations) | 2 (2) | 0 (0)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Bradycardia neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 2 (2)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 1 (1) | 2 (2)
Interleukin level increased (Investigations) | 1 (1) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 14 (14)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital pneumonia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Ureaplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCT/LCT/FO-containing 20% Fat Emulsion (N=24) | MCT/LCT Emulsion (20%) (N=24)
Anemia neonatal (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bradycardia neonatal (Cardiac disorders) | 20 (20) | 17 (17)
Congenital methemoglobinemia (Congenital, familial and genetic disorders) | 12 (12) | 13 (13)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infusion site erythema (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (4)
Amniotic infection syndrome of Blane (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 2 (2) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Base excess increased (Investigations) | 3 (3) | 1 (1)
Bilirubin conjugated increased (Investigations) | 11 (11) | 13 (13)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 24 (24) | 22 (22)
Blood lactic acid increased (Investigations) | 15 (15) | 16 (16)
Blood triglycerides increased (Investigations) | 5 (5) | 8 (8)
Body temperature increased (Investigations) | 3 (3) | 1 (1)
C-reactive protein increased (Investigations) | 5 (5) | 5 (5)
Hemoglobin decreased (Investigations) | 7 (7) | 6 (6)
Interleukin level increased (Investigations) | 19 (19) | 18 (18)
Oxygen saturation decreased (Investigations) | 5 (5) | 2 (2)
Platelet count decreased (Investigations) | 8 (8) | 8 (8)
Prothrombin level decreased (Investigations) | 2 (2) | 0 (0)
Prothrombin level increased (Investigations) | 4 (4) | 6 (6)
Red blood cell count decreased (Investigations) | 11 (11) | 15 (15)
Reticulocyte count increased (Investigations) | 15 (15) | 15 (15)
White blood cell analysis decreased (Investigations) | 8 (8) | 7 (7)
White blood cell analysis increased (Investigations) | 4 (4) | 3 (3)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 18 (18) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less